CLINICAL TRIAL: NCT05096013
Title: Effect of Individual Nutritional Therapy in Patients at Risk for Malnutrition and Sarcopenia in Pulmonary Rehabilitation - a Randomized Controlled Trial
Brief Title: Nutritional Therapy in Patients at Risk for Malnutrition and Sarcopenia in Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thimo Marcin (Other)
Collaborators: Bern University of Applied Sciences (Other)
Responsible Party: Sponsor-Investigator, Thimo Marcin, Head of Reseach Department, Berner Reha Zentrum AG
Organization: Berner Reha Zentrum AG (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-01824
Record Dates: First submitted 2021-10-05; First posted 2021-10-27 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Sarcopenia; Malnutrition
Keywords: individual nutrition therapy
MeSH Terms: conditions — Sarcopenia; Malnutrition

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Patients cannot be blinded due to the nature of the intervention. However, the personnel involved will be blinded to the collection of the primary endpoint. In order to be able to blind the nutritional calculations of the primary endpoint, the logged amounts of food eaten will be recorded on the neutral eating cards, on which the study group allocation will not be apparent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individual nutrition therapy (Experimental): Individualized nutrition therapy: Specialists in nutritional counseling determine the patient's individual energy and protein needs and create targeted individual measures to achieve them. Measures can include, for example, adjustments to the menu, food enrichment or supplementation. The measures are discussed with the patients on an ongoing basis and adjusted as necessary.
  Interventions: Other: individual nutritional therapy
- usual care (No Intervention): Usual care: Participants in the control group receive a standardized food fortification of the soups with fat and protein, as well as an energy- and protein-rich dessert. No additional advice or adjustments are made by the iNT.

INTERVENTIONS:
Other: individual nutritional therapy — Intervention arm: Usual care + individualized nutritional therapy. Patients at risk for malnutrition and sarcopenia will receive a counselling by the nutritional therapist twice a week. The therapists will assess the patient's energy and protein demand in order to develope appropriate individual measures (e.g additional meals or supplements) to increase patients' energy and protein intake. Individual nutritional therapy is already usual care in patients with high risk for malnutrition, but not for patients with only light to moderate risk of malnutrition and risk of sarcopenia.
  Arms: individual nutrition therapy

SUMMARY:
Malnutrition and sarcopenia (muscle wasting) are common in health care settings and represent a health and economic burden due to associated increased mortality and prolonged hospital stays. Nutritional therapy co-management is recommended for both diagnoses.

This study investigates the efficacy of individualized nutrition therapy (iNT) in pulmonary rehabilitation. Patients at significant risk for malnutrition already receive iNT within clinical routine during rehabilitation. The investigators will investigate if patients with only mild to moderate risk of malnutrition and possible sarcopenia also benefit from iNT.

DETAILED DESCRIPTION:
The participating patients are randomly assigned to two groups after giving written consent.

The intervention group receives individual counseling by nutrition therapists twice a week in addition to the usual rehabilitation program. The iNT determines the energy and protein needs of the patients and creates targeted individual measures to achieve them. Measures may include, for example, adjustments to the meal plan or nutritional supplementation. The measures are continuously adapted to the patients' needs.

The control group also receives soup fortified with a standard amount of protein and fat and, if needed, an energy- and protein-rich dessert option as part of the rehabilitation routine care for patients at risk for malnutrition. However, patients from the control group do not receive additional counseling or adjustment by the iNT.

Patients' energy and protein intake will be recorded on three subsequent days at start of rehabilitation and at three subsequent days before discharge. Average duration of rehabilitation is expected to be three weeks. As primary outcome, change in energy intake will be compared between groups. Additionally, change in protein intake and other follow-up parameters of nutritional status and sarcopenia will be examined.

ELIGIBILITY:
Inclusion Criteria:

* admission to rehab due to chronic obstructive pulmonary disease or after a pneumonia
* light to moderate risk of malnutrition (Nutritional Risk Score-2002: 3-4 Points)
* risk of sarcopenia (sarc-f >=4)
* signed informed consent

Exclusion Criteria:

* medically described nutritional support
* reasons (cognitive, language) that prevent a informed consent
* enteral or parenteral nutrition
* after bariatric surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Energy intake | From admission to discharge (2-3 weeks)
  Change in energy intake [kcal] from start to end of rehabilitation.

SECONDARY OUTCOMES:
protein intake | From admission to discharge (2-3 weeks)
  Change in protein intake [g] from start to end of rehabilitation.
grip strength | From admission to discharge (2-3 weeks)
  Change in grip strength (muscle strength) from start to end of rehabilitation.
lean body mass | From admission to discharge (2-3 weeks)
  Change in lean body mass (muscle mass) from start to end of rehabilitation.
time up and go | From admission to discharge (2-3 weeks)
  Change in time up an go time (muscle function) from start to end of rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Berner Reha Zentrum, Heiligenschwendi, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2022, July

REFERENCES:
- [Derived] Coiro M, Zurfluh A, Lehmann U, Brun P, Scheel-Sailer A, Tschanz H, van Hoof A, Wilhelm M, Marcin T. Effect of individual nutritional therapy during inpatient pulmonary rehabilitation in patients at risk for malnutrition and sarcopenia - a randomized controlled trial. Chron Respir Dis. 2025 Jan-Dec;22:14799731251350692. doi: 10.1177/14799731251350692. Epub 2025 Jun 15. PMID 40518743